CLINICAL TRIAL: NCT00269919
Title: Effect on Efficacy, Safety and Quality of Life by Long-Term Treatment of Long-Acting Risperidone Microspheres in Patients With Schizophrenia
Brief Title: An Efficacy and Safety Study of Long-Term Risperidone Microspheres in Participants With Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR002089; RIS-KOR-64
Record Dates: First submitted 2005-12-22; First posted 2005-12-26 (Estimated); Results first posted 2013-08-09 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-03

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia; Risperidone; Risperidal Consta
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Risperidone Long-Acting Injectable (RLAI) (Experimental): The RLAI 25 milligram (mg) or 37.5 mg or 50 mg will be administered intramuscularly (into a muscle) depending on Investigator's discretion every 2 weeks for 2 years.
  Interventions: Drug: Risperidone Long-Acting Injectable (RLAI)

INTERVENTIONS:
Drug: Risperidone Long-Acting Injectable (RLAI) — The RLAI 25 mg or 37.5 mg or 50 mg will be administered intramuscularly depending on Investigator's discretion every 2 weeks for 2 years.

SUMMARY:
The purpose of this study is to evaluate the long-term efficacy and safety of a long-acting injectable formulation of risperidone (an antipsychotic medication) and its influence on quality of life, in participants with schizophrenia (psychiatric disorder with symptoms of emotional instability, detachment from reality, often with delusions and hallucinations, and withdrawal into the self).

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention) single-arm, and prospective study (study following participants forward in time) of risperidone microspheres in participants with schizophrenia. Participants will be treated with intramuscular (into a muscle) injections of either 25 milligram (mg) or 37.5 mg or 50 mg of risperidone twice weekly, every 2 weeks for 2 years. The total duration of study will be 2 years. The efficacy of participants will primarily be evaluated by total Positive and Negative Syndrome Scale (PANSS) score. Participants' quality of life and safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with schizophrenia or schizoaffective disorder (in-patients or out-patients)
* Participants currently having their symptoms well controlled with a stable dose of oral antipsychotic medication
* Participants who have signed informed consent form Exclusion Criteria:
* Participants who have never received any previous antipsychotic treatment
* Participants who have received clozapine during the last 3 months
* Participants with a serious unstable medical condition, including laboratory abnormalities
* Participants with a history of, or current symptoms of tardive dyskinesia (a complication of neuroleptic therapy involving involuntary movements of facial muscles) or neuroleptic malignant syndrome (a rare psychotropic-drug reaction, which may be characterized by confusion, reduced consciousness, high fever or pronounced muscle stiffness)
* Female participants who are pregnant or breast-feeding, or are of childbearing age without adequate contraception

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-08; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd., Korea Clinical Trial, Study Director — Janssen Korea, Ltd., Korea
Locations (1):
- Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Groups:
- Risperidone Long-acting Injection (RLAI): The RLAI 25 milligram (mg) or 37.5 mg or 50 mg was administered intramuscularly (into a muscle) depending on Investigator's discretion every 2 weeks for 2 years.
Period: Overall Study
Arm/Group | Risperidone Long-acting Injection (RLAI)
Started | 40
Treated | 39
Completed | 13
Not Completed | 27
Not completed — Other | 26
Not completed — Started but not treated | 1

BASELINE CHARACTERISTICS:
Groups:
- Risperidone Long-acting Injection (RLAI): The RLAI 25 milligram (mg) or 37.5 mg or 50 mg was administered intramuscularly depending on Investigator's discretion every 2 weeks for 2 years.
Arm/Group | Risperidone Long-acting Injection (RLAI)
Number analyzed (Participants) | 39
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.0 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 25

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Positive and Negative Syndrome Scale (PANSS) Score at Week 96
Description: The PANSS is a 30-item scale consisting of 3 subscales, the positive subscale (7 items), the negative subscale (7 items), and the general psychopathology subscale (16 items) and it is designed to assess various symptoms of schizophrenia including delusions, grandiosity, blunted affect, poor attention, and poor impulse control. The 30 items are rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme). The PANSS total score consists of the sum of all 30 PANSS items and ranges from 30 (absent) to 210 (extreme ill). Higher scores indicate worsening.
Time Frame: Baseline and Week 96
Population: The intent-to-treat (ITT) analysis population included all the participants who received at least 1 dose of study medication, satisfied all the eligibility criteria and provided at least 1 efficacy measurement post-baseline. Here, 'N'=the participants who were evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Risperidone Long-Acting Injection (RLAI)
Number analyzed (Participants) | 37
Units on a scale
  Baseline | 73.00 (13.98)
  Change at Week 96 | 18.24 (14.87)

2. Secondary Outcome: Change From Baseline in Clinical Global Impression-Severity (CGI-S) Score at Week 96
Description: The CGI-S rating scale is used to rate the severity of a participant's psychotic condition on a 7-point scale. It is rated as follows: 1=Normal, not at all ill, 2=Borderline mentally ill, 3=Mildly ill, 4=Moderately ill, 5=Markedly ill, 6=Severely ill, and 7=Among the most extremely ill. Higher scores indicate worsening.
Time Frame: Baseline and Week 96
Population: The ITT analysis population included all the participants who received at least 1 dose of study medication, satisfied all the eligibility criteria and provided at least 1 post-baseline efficacy measurement. Here, 'N'=the participants who were evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Risperidone Long-Acting Injection (RLAI)
Number analyzed (Participants) | 37
Units on a scale
  Baseline | 4.62 (0.68)
  Change at Week 96 | -0.89 (1.15)

3. Secondary Outcome: Change From Baseline in Global Assessment of Functioning (GAF) Score at Week 96
Description: GAF is a 100-point tool rating overall psychological, social and occupational functioning of adults. The higher score range (91-100) refers to a superior functioning in a wide range of activities, and absence of symptoms. The lower score range (1-10) refers to persistent danger of severely hurting self or others; or persistent inability to maintain minimum personal hygiene; or serious suicidal act with clear expectation of death. Lower scores indicate worsening.
Time Frame: Baseline and Week 96
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Risperidone Long-Acting Injection (RLAI)
Number analyzed (Participants) | 37
Units on a scale
  Baseline | 44.32 (12.21)
  Change at Week 96 | 8.86 (15.80)

4. Secondary Outcome: Change From Baseline in World Health Organization (WHO)-Quality of Life (QOL) at Week 96
Description: The WHOQOL-BREF is a 26-item, self-report questionnaire and short version of WHOQOL-100, consisting of 4 domains: physical health (7 items), psychological health (6 items), social relationships (3 items), and environmental health (8 items); it also contains QOL and general health items. Domain scores are scaled in a positive direction (i.e. higher scores denote higher quality of life). The mean score of items within each domain is used to calculate the domain score. Each individual item of the WHOQOL-BREF is scored from 1=not at all to 5=completely on a response scale, which is stipulated as a 5-point ordinal scale. The scores are then transformed linearly to a scale of 0 (the worse quality of life) to 100 (the worse quality of life).
Time Frame: Baseline and Week 96
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Risperidone Long-Acting Injection (RLAI)
Number analyzed (Participants) | 36
Units on a scale
  Baseline | 71.22 (15.79)
  Change at Week 96 | 2.06 (15.85)

5. Secondary Outcome: Change From Baseline in Neurocognitive Function Test (NCFT): General Intelligence (Korean-Wechsler Adults Intelligence Scale [K-WAIS]) at Week 96
Description: The K-WAIS is a Korean version of the Wechsler Adult Intelligence Scale-Revised (WAIS-R). It is an intelligence test that assess 3 general areas of intelligence quotients (IQ): verbal IQ, performance IQ and full-scale IQ (FSIQ). The verbal IQ includes: Digit Span, Vocabulary, and Arithmetic; performance IQ includes: Picture Arrangement and Block Design; and FSIQ is an IQ assessed by measuring an individual's overall level of general cognitive and intellectual functioning. The highest FSIQ is 160. The greater the quotient, higher the level of intelligence.
Time Frame: Baseline and Week 96
Population: The ITT analysis population included all participants who received at least 1 dose of study medication, satisfied all eligibility criteria and provided at least 1 post-baseline efficacy measurement. Here 'N'=participants who were evaluated for this outcome measure and 'n'=participants who were evaluated for this outcome measure at given time point.
Measure: Mean (Standard Deviation); unit: Intelligence quotient (IQ)
Arm/Group | Risperidone Long-Acting Injection (RLAI)
Number analyzed (Participants) | 29
Intelligence quotient (IQ)
  Baseline: GI, Digit Span (n=28) | 11.39 (2.35)
  Change at Week 96: GI, Digit span (n=28) | 1.36 (1.63)
  Baseline: GI, Vocabulary (n=29) | 12.28 (3.12)
  Change at Week 96: GI, Vocabulary (n=29) | 1.18 (1.33)
  Baseline: GI, Arithmetic (n=29) | 10.00 (2.38)
  Change at Week 96: GI, Arithmetic (n=29) | 1.18 (2.18)
  Baseline: GI, Picture arrange (n=29) | 10.10 (2.68)
  Change at Week 96: GI, Picture arrange (n=29) | 2.36 (3.07)
  Baseline: GI, Block Design (n=29) | 11.59 (2.44)
  Change at Week 96: GI, Block Design (n=29) | 0.82 (2.23)
  Baseline: GI, FSIQ (n=29) | 106.07 (15.32)
  Change at Week 96: GI, FSIQ (n=29) | 10.64 (11.98)

6. Secondary Outcome: Change From Baseline in NCFT: Controlled Oral Word Association Test at Week 96
Description: The Controlled Oral Word Associated Test is a measure of verbal fluency, which requires participants to generate words orally that begin with a given letter of the alphabet. Participants are given 1 min to name as many words as possible. Performance was calculated by the number of words generated in the 1-min period. This measure, requiring rapid and organized word retrieval, is a sensitive indicator of brain dysfunction.
Time Frame: Baseline and Week 96
Population: The ITT analysis population included all participants who received at least 1 dose of study medication, satisfied all eligibility criteria and provided at least 1 post-baseline efficacy measurement. Here 'N'=participants who were evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: Words generated per min
Arm/Group | Risperidone Long-Acting Injection (RLAI)
Number analyzed (Participants) | 28
Words generated per min
  Baseline: corrected response | 10.25 (2.61)
  Change at Week 96: corrected response | 0.00 (1.83)

7. Secondary Outcome: Change From Baseline in NCFT: Rey Kim Memory Test-Korean Auditory Verbal Learning Test (KAVLT) at Week 96
Description: The KAVLT is a neuropsychological assessment designed to evaluate verbal memory in participants. The KAVLT is useful in evaluating the nature and severity of memory dysfunction and to track changes in memory function over time. The test is designed as a list-learning paradigm in which the participants hears a list of 15 words, and are asked to recall as many words from the list as possible. This procedure is carried out a total of 5 times. Then a second list of 15 words is presented, allowing the participants only 1 attempt to recall. Immediately following this, the participants are asked to remember as many words as possible from the first list. KAVLT consists of 2 test conditions: Delayed Recall and Delayed Recognition. The upper limit for 'words recalled' is 15, which represents better episodic memory.
Time Frame: Baseline and Week 96
Population: The ITT analysis population included all participants who received at least 1 dose of study medication, satisfied all eligibility criteria and provided at least 1 post-baseline efficacy measurement.Here 'N'=participants who were evaluated for this outcome measure and 'n'=participants who were evaluated for this outcome measure at given time point.
Measure: Mean (Standard Deviation); unit: Words recalled
Arm/Group | Risperidone Long-Acting Injection (RLAI)
Number analyzed (Participants) | 28
Words recalled
  Baseline: Trial 1 (n=27) | 9.81 (3.50)
  Change at Week 96: Trial 1 (n=27) | 2.30 (1.89)
  Baseline: Trial 2 (n=28) | 8.71 (3.10)
  Change at Week 96: Trial 2 (n=28) | 1.60 (3.34)
  Baseline: Trial 3 (n=28) | 7.96 (4.39)
  Change at Week 96: Trial 3 (n=28) | 2.40 (3.10)
  Baseline: Trial 4 (n=28) | 8.39 (3.92)
  Change at Week 96: Trial 4 (n=28) | 0.90 (3.63)
  Baseline: Trial 5 (n=28) | 8.50 (3.84)
  Change at Week 96: Trial 5 (n=28) | 1.50 (2.22)
  Baseline: delayed recall (n=28) | 8.50 (3.96)
  Change at Week 96: delayed recall (n=28) | 2.90 (4.65)
  Baseline: delayed recognition (n=28) | 9.21 (2.63)
  Change at Week 96: delayed recognition (n=28) | 1.50 (3.72)

8. Secondary Outcome: Change From Baseline in NCFT: Rey Kim Memory Test- Korean-Rey Complex Figure Test (K-RCFT) at Week 96
Description: The RCFT is a neuropsychological assessment designed to evaluate visual memory in participants. The RCFT is useful in evaluating the spatial perception and visual memory. The RCFT consists of 3 test conditions: Copy, Immediate Recall and Delayed Recall. At the first step, participants are given the RCFT stimulus card, and then asked to draw the same figure. Subsequently, they are instructed to draw what they remembered. Then, after a delay of 30 min, they are required to draw the same figure once again, a score of 2 points for each drawn element (a complete straight line or a circle) remembered correctly. The total score is the sum of points scored for each correctly drawn element and it ranges from 0 to 36. The maximum score indicates excellent visual memory.
Time Frame: Baseline and Week 96
Population: The ITT analysis population included all participants who received at least 1 dose of study medication, satisfied all eligibility criteria and provided at least 1 post-baseline efficacy measurement.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Risperidone Long-Acting Injection (RLAI)
Number analyzed (Participants) | 28
Units on a scale
  Baseline: copy | 15.11 (1.40)
  Change at Week 96: copy | -0.10 (1.91)
  Baseline: immediate recall | 8.75 (4.44)
  Change at Week 96: immediate recall | 2.20 (3.85)
  Baseline: delayed recall | 9.18 (3.43)
  Change at Week 96: delayed recall | 1.70 (2.50)

9. Secondary Outcome: Change From Baseline in NCFT: Memory Quotient (MQ) at Week 96
Description: MQ was obtained by adding up the results of verbal memory and visual memory test. The memory quotient will include learning curve, memory retention, retrieval efficiency, drawing/memory consistency, verbal/visual memory consistency and intelligence/memory consistency. The highest MQ is 160, which indicates excellent memory.
Time Frame: Baseline and Week 96
Population: The ITT analysis population included all participants who received at least 1 dose of study medication, satisfied all eligibility criteria and provided at least 1 post-baseline efficacy measurement. Here, "N" is the number of participants evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: MQ
Arm/Group | Risperidone Long-Acting Injection (RLAI)
Number analyzed (Participants) | 28
MQ
  Baseline | 93.71 (15.07)
  Change at Week 96 | 10.70 (12.58)

10. Secondary Outcome: Change From Baseline in NCFT: Trail Making Test (TMT)-Time at Week 96
Description: TMT is attention, mental flexibility, visual search, motor function measure test. Test is divided into A and B types. Participants using a pencil or connect numbers in sequence (A-type), in turn, alternating between numbers and letters must be connected (B-type). The test measures the response time.
Time Frame: Baseline and Week 96
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Risperidone Long-Acting Injection (RLAI)
Number analyzed (Participants) | 29
Seconds
  Baseline: Trail A-time | 39.83 (14.95)
  Change at Week 96: Trail A-time | -3.18 (10.48)
  Baseline: Trail B-time | 96.03 (33.31)
  Change at Week 96: Trail B-time | -16.0 (32.49)

11. Secondary Outcome: Change From Baseline in NCFT: TMT-Error at Week 96
Description: TMT is attention, mental flexibility, visual search, motor function measure test. Test is divided into A and B types. Participants using a pencil or connect numbers in sequence (A-type), in turn, alternating between numbers and letters must be connected (B-type). The test measures the the number of errors.
Time Frame: Baseline and Week 96
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Errors
Arm/Group | Risperidone Long-Acting Injection (RLAI)
Number analyzed (Participants) | 28
Errors
  Baseline: Trail A-error | 0.11 (0.31)
  Change at Week 96: Trail A-error | 0.00 (0.50)
  Baseline: Trail B-error | 0.68 (1.28)
  Change at Week 96: Trail B-error | -1.11 (2.42)

12. Secondary Outcome: Liverpool University Neuroleptic Side Effect Rating Scale (LUNSERS) Score
Description: The LUNSERS is a self-report measure of antipsychotic side effects. It consists of 51 questions, 41 questions on side effects and 10 questions are of "red herrings" to validate the results. Each question is rated on a 4-point scale, where 0=not at all; and 4=very much. The total neuroleptic side effect score is the sum of the scores for the side effects items (i.e. all items excluding the red herrings). Total side effects score ranges from 0 to 164, where 0 to 40=low side effect rating, 41 to 80=medium side effect rating and greater than 81=high side effect rating.
Time Frame: Baseline and Week 96
Population: The safety analysis population included all the participants who participated in the clinical trial and received at least 1 dose of RLAI. Here, 'N'=the participants who were evaluated for this outcome measure and 'n'=the participants who were evaluated for this outcome measure at given time point.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Groups:
- Risperidone Long-Acting Injection (RLAI): The RLAI 25 milligram (mg) or 37.5 mg or 50 mg had been administered intramuscularly depending on Investigator's discretion every 2 weeks for 2 years.
Arm/Group | Risperidone Long-Acting Injection (RLAI)
Number analyzed (Participants) | 38
Unit on a scale
  Baseline | 101.32 (39.90)
  Week 96 (n=13) | 76.54 (17.34)

13. Secondary Outcome: Change From Baseline in Drug Attitude Inventory-10 (DAI-10) Item Scale Score at Week 96
Description: The DAI-10 is a 10-item questionnaire to assess 1) subjective experience of medication and 2) attitudes and beliefs toward neuroleptics which may influence medication compliance in schizophrenia participants. It is the binary scale assessing the participant's subjective response. A 'compliant' response is scored as +1; a dysphoric response is scored as -1. A positive sum of items indicates a positive subjective response (SR); a negative sum of scores indicates a negative SR (non-compliant). The final score for each person at each time is the positive score minus the negative score.
Time Frame: Baseline and Week 96
Population: The ITT analysis population included all the participants who received at least 1 dose of study medication, satisfied the eligibility criteria and provided at least 1 post-baseline efficacy measurement. Here, 'N'=the participants who were evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Risperidone Long-Acting Injection (RLAI)
Number analyzed (Participants) | 36
Units on a scale
  Baseline | -0.22 (4.92)
  Change at Week 96 | 0.28 (4.51)

14. Secondary Outcome: Total Drug Induced Extra-Pyramidal Symptoms Scale (DIEPSS) Score
Description: A scale used to assess the extrapyramidal symptoms attributable to antipsychotics. It consists of 9 items (8 to assess individual symptoms and 1 to assess global severity). Each item is assessed from 0 (none, normal) to 4 (severe). The total score is the sum of the 8 item scores, for a total range of 0 (normal) to 32 (severe). The items for the assessment of individual symptoms are classified into 4 categories of parkinsonism, akathisia, dystonia and dyskinesia.
Time Frame: Baseline and Week 96
Population: The safety analysis population included all the participants who participated in the clinical trial and received at least 1 dose of risperidone long acting injection (RLAI). Here, 'N'=the participants who were evaluated for this outcome measure and 'n'=the participants who were evaluated for this outcome measure at given time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Risperidone Long-Acting Injection (RLAI)
Number analyzed (Participants) | 38
Units on a scale
  Baseline | 4.13 (1.12)
  Week 96 (n=12) | 2.50 (1.45)

ADVERSE EVENTS:
Time Frame: Baseline up to 2 years
Arm/Group | Risperidone Long-acting Injection (RLAI)
Serious Adverse Events (participants affected / at risk) | 6/39
Other Adverse Events (participants affected / at risk) | 27/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Risperidone Long-acting Injection (RLAI) (N=39)
Schizophrenia (Psychiatric disorders) | 2
Psychotic disorder (Psychiatric disorders) | 3
Cardiac disorders (Cardiac disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Risperidone Long-acting Injection (RLAI) (N=39)
Akathisia (Nervous system disorders) | 5
Headache (Nervous system disorders) | 3
Oral pain (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 2
constipation (Gastrointestinal disorders) | 2
Upper respiratory tract infection (Infections and infestations) | 8
Insomnia (Psychiatric disorders) | 3
Vision blurred (Eye disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 2
Amenorrhea (Reproductive system and breast disorders) | 2

LIMITATIONS AND CAVEATS:
There is limitation in the study that selection or observer bias may occur because this clinical trial was an open, non-comparative, single-arm study and precaution would be necessary for interpreting change in various scales observed in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less